CLINICAL TRIAL: NCT05731622
Title: Effect of a Single Instillation of Mitomycin C on the Intravesical Recurrence Rate After Ureteroscopy for Upper Tract Urothelial Carcinoma: A Prospective, Multicenter Study
Brief Title: Effect of a SI-MMC on the IVR Rate After Ureteroscopy for UTUC
Acronym: SINCERE
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Joyce Baard, drs J. Baard Urologist (PI), Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W22_369
Record Dates: First submitted 2023-01-24; First posted 2023-02-16 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Upper Urinary Tract Carcinoma
Keywords: Intravesical recurrence; Mitomycin C; Ureteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the intravesical recurrence (IVR) rate after ureteroscopy (diagnostic or treatment) for upper tract urothelial carcinoma (UTUC) followed by an adjuvant single instillation of Mitomycin C (SI-MMC).

The main question it aims to answer are:

* What is the total and time to IVR after 2 years after ureteroscopy (diagnostic or treatment) for UTUC
* How is the IVR compared with a historical cohort (no SI-MMC)
* What is the time to IVR after 2 years in patients who subsequently received treatment by endoscopy vs. radical nephroureterectomy (RNU)
* What is the additional value of a SI-MMC on time to IVR after RNU + adjuvant MMC in patients who were evaluated by ureteroscopy prior to RNU

DETAILED DESCRIPTION:
The primary objective is to evaluate the IVR rate after ureteroscopy (diagnostic or treatment) followed by an single instillation of MMC (SI-MMC), in patients with clinically non-metastatic UTUC.

The main question we aim to answer are:

* What is the total and time to IVR after 2 years after ureteroscopy (diagnostic or treatment) for UTUC
* How is the IVR compared with a historical cohort (no SI-MMC)
* What is the time to IVR after 2 years in patients who subsequently received treatment by endoscopy vs. radical nephroureterectomy
* What is the additional value of a SI-MMC on time to IVR after RNU + adjuvant MMC in patients who were evaluated by ureteroscopy prior to RNU.

Secondary objectives include the evaluation of possible predictive factors for IVR rate.

Study design: Multicentre, prospective cohort study in a clinical setting,

Study population: All adult patients (age ≥18 years) with a (suspicion of a) urothelial carcinoma of the upper urinary tract undergoing ureteroscopy, either diagnostic or as endoscopic kidney sparing treatment, followed by a post-operative single instillation of Mitomycin C.

Intervention: No intervention

Main study parameters/endpoints:

The primary endpoint of this study is the time to and total intravesical recurrences (histological proven) in the first 24 months following ureteroscopy (diagnostic or treatment) for UTUC followed a single instillation of Mitomycin C.

Secondary Objective(s): to evaluate possible predictive factors for IVR rate looking at gender, tumour size, tumour focality, tumour location, postoperative stent placement, use of an ureteral access sheath, timing of administration of MMC, the performance of an endoscopic biopsy during ureteroscopy.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Investigations during follow-up include cystoscopy, ureteroscopy and CT-urography, which is in line with the standardized care and will not include additional investigations.

ELIGIBILITY:
Inclusion Criteria:

* All patients suspect for having non-metastatic disease and planned for ureteroscopy (diagnostic or treatment) and adjuvant single instillation of Mitomycin C
* Age ≥18 years
* Written informed consent

Exclusion Criteria:

* History of histological proven urothelial carcinoma of the bladder, including carcinoma in situ
* History of histological proven UTUC in the contralateral kidney
* Concurrent bladder tumour found pre-operatively or per-operatively
* Patients where it is not feasible to obtain histology by biopsies intra-operatively
* Known Mitomycin C
* Renal transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspect of having non-metastatic UTUC
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Time to and total number of Intravesical recurrences (IVR) | 2 years
  What is the time to and total number of IVR 2 years after ureteroscopy (diagnostic or treatment) with SI-MMC for UTUC
Time to and total number of IVR after endoscopic vs radical treatment | 2 years
  What is the time to and total number of IVR after 2 years in patients who subsequently received treatment by endoscopy vs. radical nephroureterectomy
Time to and total IVR after diagnostic ureteroscopy in patients who received final treatment by RNU | 2 years
  Is there an additional value of SI-MMC on total and time to IVR after RNU in patients who were evaluated by ureteroscopy prior to RNU. Outcome measurement (time to IVR and total IVR) will be compared to a historical cohort who did not receive Mitomycin C to evaluate the additional effect

SECONDARY OUTCOMES:
predictive factors for IVR | 2 years
  to evaluate possible predictive factors for IVR rate looking different variables by multivariate logistic regression; with the dependent variable IVR and independent variables: gender (male/ female), tumour size (< 2cm/ >2cm), tumour focality (unifocal/ multifocal), tumour invasiveness (invasive/ non-invasive), tumour location (ureter/ puelocaliceal), use of Urethral access sheath (yes/no), use of postoperative stent (yes/ no), timing of MMC administartion (<24h/>24h)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Baard, MD, MSc, Principal Investigator — AmsterdamUMC
Locations (1):
- AmsterdamUMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided